CLINICAL TRIAL: NCT06040528
Title: Barts Early Post-Acute Myocardial Infarction Discharge Registry
Brief Title: Early Discharge Pathway Registry
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: AWAIT
Record Dates: First submitted 2022-12-22; First posted 2023-09-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevation Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients discharged on the Early Discharge Pathway at Barts Heart Centre: This study aims to assess, in a real-world setting, the safety, efficacy and feasibility of further investigations in patients with acute coronary syndrome who are admitted to Barts Heart Centre and are discharged via the early discharge pathway.

SUMMARY:
Despite the year-on-year decrease, coronary artery disease (CAD) still remains one of the leading causes of mortality worldwide. With advances in technology and our understanding of cardiac disease, we can now treat CAD using minimally invasive interventional techniques. This has revolutionised treatment for and improved the lives of many patients with CAD. Although trials have assessed various therapeutic strategies in various populations, real-world evidence of intervention and medical treatment among patients with CAD is increasingly recognised as an important part of providing safety and efficacy data and improving the care we provide.

Regional heart attack services have improved clinical outcomes following ST-segment elevation myocardial infarction (STEMI) by facilitating early reperfusion by primary percutaneous coronary intervention (PCI). Early discharge after primary PCI is welcomed by patients and increases the efficiency of health care.

This data will add to that literature by assessing the characteristics and outcomes of patients with CAD, concentrating on those who are discharged via the early discharge pathway. It will also identify and characterise predictors of outcomes, and improve risk stratification and diagnostic evaluation.

DETAILED DESCRIPTION:
The proposed study includes one of the largest coronary interventional programmes in the UK at Europe's largest cardiac centre (BHC). This has allowed us to accumulate a large number of patients in just over 4 years. All patients admitted with acute coronary syndrome and discharged via the early discharge pathway are included in this study using a clinical database. The database is password-protected and includes demographic, clinical and outcome data.

The database includes patients with simple to complex CAD. We will use this database to test several hypotheses including but not limited to investigating characteristics of patients treated, complications of interventional treatment and outcomes of patients. This research will add substantially to the literature by providing real-world data from a leading coronary centre.

In this registry, we will assess the safety and feasibility of the EHD pathway for patients who were discharged after primary PCI from a high-volume heart attack centre in London.

The impact of this study will have local, regional and global consequences with an emphasis on investigating poorly studied areas (e.g. decompensated aortic stenosis) and providing evidence to improve their management and stimulate further research.

ELIGIBILITY:
Inclusion Criteria:

Informed consent will not be sought for, as patients are automatically included onto a database that we will use for research purposes. No children will be included in this study. Vulnerable adults or those unable to give consent will be included in the study as well if they are referred to the Interventional Cardiology team.

Both male and female patients ≥16 years of age will be included

All patients will have been admitted to BHC with acute coronary syndrome.

Exclusion Criteria:

Patients <16 years will not be included in this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include all patients admitted to or reviewed at Barts Heart Centre (St. Bartholomew's Hospital) who are discharged via the early discharge pathway. These patients range from young adults to the elderly and will include any patient ≥16 years of age. Patients who are followed up with and without any intervention (i.e. both medically managed patients as well as patients undergoing intervention) are equally as important and therefore we shall include both groups of patients.
  Patients will be included from referrals made by other clinicians either as in or outpatients. All these patients have their clinical data captured on a database or hospital based clinical programme.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of Titration of medication | 1 year
  To assess how medical therapy has been titrated in patients on the early discharge pathway
Measurement of MACE | 1 year
  Assessment of MACE events in patients on the early discharge pathway
Assessment of Quality of Life | 1 year
  Assess QoL using Questionnaire to assess change in symptoms at 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Barts Health NHS Trust, London
  - Dr. Daniel Jones, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones DA, Rathod KS, Howard JP, Gallagher S, Antoniou S, De Palma R, Guttmann O, Cliffe S, Colley J, Butler J, Ferguson E, Mohiddin S, Kapur A, Knight CJ, Jain AK, Rothman MT, Mathur A, Timmis AD, Smith EJ, Wragg A. Safety and feasibility of hospital discharge 2 days following primary percutaneous intervention for ST-segment elevation myocardial infarction. Heart. 2012 Dec;98(23):1722-7. doi: 10.1136/heartjnl-2012-302414. Epub 2012 Oct 10. PMID 23053711
- [Background] Jones DA, Rathod KS, Mathur A, Archbold RA. Discharge after primary percutaneous coronary intervention: the earlier the better? Eur Heart J Qual Care Clin Outcomes. 2022 May 5;8(3):229-231. doi: 10.1093/ehjqcco/qcab100. No abstract available. PMID 34951919
- [Background] Rathod KS, Comer K, Casey-Gillman O, Moore L, Mills G, Ferguson G, Antoniou S, Patel R, Fhadil S, Damani T, Wright P, Ozkor M, Das D, Guttmann OP, Baumbach A, Archbold RA, Wragg A, Jain AK, Choudry FA, Mathur A, Jones DA. Early Hospital Discharge Following PCI for Patients With STEMI. J Am Coll Cardiol. 2021 Dec 21;78(25):2550-2560. doi: 10.1016/j.jacc.2021.09.1379. PMID 34915986